CLINICAL TRIAL: NCT05291676
Title: Systems Investigation of Vaccine Responses in Aging and Frailty
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000035834; U19AI089992 (NIH); 0409027018 (Other: previous Yale IRB)
Record Dates: First submitted 2022-03-07; First posted 2022-03-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Influenza
Keywords: vaccine; influenza vaccine; older adults; vaccine response; toll-like receptors; immune response
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluad vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 21-30 standard dose Fluad (Active Comparator): Participants age 21-30 years will receive the standard dose Fluad
  Interventions: Biological: Fluad
- 21-30 high dose Fluzone (Active Comparator): Participants age 21-30 years will receive the high dose Fluzone
  Interventions: Biological: Fluzone
- ≥65 years standard dose Fluad (Experimental): Participants age ≥65 years will receive standard dose Fluad
  Interventions: Biological: Fluad
- ≥65 years high dose Fluzone (Experimental): Participants age ≥65 years will receive high dose Fluzone
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluzone — Fluzone High-Dose 0.7 ml intramuscular injection, standard as recommended by manufacturer
  Arms: 21-30 high dose Fluzone; ≥65 years high dose Fluzone
Biological: Fluad — Fluad Quadrivalent, MF59 adjuvanted 0.5 ml intramuscular injection, standard as recommended by manufacturer
  Arms: 21-30 standard dose Fluad; ≥65 years standard dose Fluad

SUMMARY:
This study will compare the immune response signatures (including immunologic, transcriptomic and metabolomic) of the two influenza vaccines approved for use in adults age 65 and over (Fluad and Fluzone High-Dose).

DETAILED DESCRIPTION:
There are two vaccines currently approved for use in adults age 65 and greater: a high-dose (HD) influenza vaccine (Fluzone High-Dose) that contains 4 times the hemagglutinin dose found in the standard vaccine, and a standard-dose (SD) vaccine containing the proprietary MF59 adjuvant (Fluad). Both vaccines give significantly highly antibody responses to influenza in older adults. This study will directly compare the HD and SD vaccines in nursing home residents, the population of older adults most vulnerable to influenza outbreaks and morbidity and mortality. It will comprehensively study the innate and adaptive response to vaccination, as well as elucidate transcriptomic and proteomic signatures of vaccine response.

This is a randomized, open label study comparing the two vaccines currently approved for use in adults age ≥ 65 years: the high-dose influenza vaccine and the MF59 adjuvanted standard-dose vaccine, both quadrivalent. The young group will be comprised of individuals 21-30 years of age, and the older cohorts will consist of nursing home residents ≥65 years. Participants will also be evaluated for evidence of influenza-like illness (ILI). ILI is defined to include clinical presentation in older adults: by the presence of either two respiratory symptoms (cough, sore throat, shortness of breath, and nasal stuffiness) or one respiratory and one systemic symptom (headache, malaise, temperature >99° F, report of feverishness and muscle aches, or altered mental status). Diagnoses of influenza will be confirmed using a real-time polymerase chain reaction (PCR) test on a nasopharyngeal (NP) swab specimen done by the hospital Virology Laboratory and facilitated by the participating medical directors.

Although this is neither an efficacy or effectiveness study, participants will be randomized 1:1 to either the high-dose influenza vaccine or the MF59 vaccine within age strata. This will ensure a non-biased allocation of the two vaccines and attempts to balance participant characteristics within age strata.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-40 or 65 and older
* Ability to understand and give informed consent (surrogate consent may apply to nursing home subjects who are decisionally impaired, with verbal assent to be obtained from subject)
* Plan to be in the New Haven, CT area for the next 4-6 weeks

Exclusion Criteria:

* Current use of medication, such as antibiotics in past two weeks. To clarify, patients taking antibiotics for the reason of a current acute infection will not be eligible. Those potential participants receiving antibiotics for prophylaxis purposes will be eligible to participate. The intention is not to create a separate group to drawn conclusions, but not to exclude these participants who are not acutely ill.
* Evidence of acute infection, identified by self- report of fever or symptoms in past two weeks
* Treatment for cancer in past three months.
* Previous adverse reaction to influenza vaccine requiring medical attention, such as allergic response (rash, anaphylaxis) or Guillain-Barré syndrome.
* Pregnant/possibly pregnant.
* History of organ, bone marrow or stem cell transplant, liver cirrhosis, kidney disease requiring dialysis, HIV/AIDS, hepatitis C or active hepatitis B
* Blood donation of 1 pint or more in past 2 months
* Treatment with clinical trial medication
* Presence of any other condition (e.g., geographical or social), actual or projected, that the investigator feels would restrict or limit the patient's participation for the duration of the study. This provision includes participants who have 50% or more missed appointments in the last three months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in production of IL-6 in monocytes to assess innate immune inflammatory response | Baseline and at Day 2, 7, and 28 post-vaccine
  Measurement of IL-6 production in monocytes via flow cytometry

SECONDARY OUTCOMES:
Change in Hemagglutination inhibition titer (HAI) in response to vaccination | Baseline and Day 28
  HAI titers levels in blood measured prior to and at day 28 post-vaccine
Change in transcriptomic analyses of gene expression | At Baseline, Day 2, Day 7, Day 28 and Day 70
  RNA-seq analysis of RNA derived from peripheral blood mononuclear cells (PBMCs) and platelet-rich plasma (PRP)
Change in proteomic analyses | At Baseline, Day 2, Day 7, Day 28 and Day 70
  Analysis of protein expression using Mass Spectrometry in plasma
Number of participants with changes in innate immune function from PBMCs and PRP as assessed using flow cytometry | At Baseline, Day 2, Day 7, Day 28 and Day 70
  Analyses will include intracellular production of cytokines including IL-10 and TNF-alpha in monocyte populations from PBMCs and expression of platelet activation markers such as CD63 and P-selectin on platelets. The effects of ex vivo Toll-like Receptor stimulation on these parameters will also be assessed.
Number of participants with changes in B and T cell function from PBMCs as assessed using flow cytometry | At Baseline, Day 2, Day 7, Day 28 and Day 70
  This will include analysis of number and proportion of antibody-secreting cells post-vaccine, and analyses of T cells following ex vivo stimulation of PBMCs with influenza hemagglutinins.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Shaw, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with Protected Health Information (PHI) removed on participant demographics and health conditions, and primary and secondary outcome data will be uploaded to the NIH ImmPort as required by the NIH Human Immunology Project Consortium.
  Publicly available data will be released after publication. Registration on ImmPort required by the NIH. Timeframe for data upload will be approximately 6-12 months after each influenza vaccine season during the study.